CLINICAL TRIAL: NCT07241468
Title: An Exploratory Clinical Study on the Safety and Efficacy of Anti-CD19/BCMA Universal Chimeric Antigen Receptor T Cells in the Treatment of Relapsed/Refractory Immune-mediated Kidney Disease
Brief Title: An Exploratory Clinical Study on the Safety and Efficacy of Anti-CD19/BCMA U CAR-T Cells in the Treatment of Relapsed/Refractory Immune-mediated Kidney Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2025-362
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Immune Nephropathy; Relapsed/Refractory Immune-mediated Kidney Disease
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/BCMA U CAR T cells (Experimental)
  Interventions: Biological: anti-CD19/BCMA U CAR T

INTERVENTIONS:
Biological: anti-CD19/BCMA U CAR T — To evaluate the safety and effectiveness of anti-CD19/BCMA CAR T cells (KN3601) in patients with immune nephropathy. All subjects will receive fludarabine/cyclophosphamide lymphodepletion followed by anti-CD19/BCMA U CAR T cells infusion.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of anti-CD19/BCMA U CAR T cell injection (KN3601) in patients with Relapsed/Refractory immune-mediated kidney disease

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old and ≤ 70 years old, male or female;
2. 2 B cell CD19 positive expression in peripheral blood detected by flow cytometry;
3. The functions of critical organs meet the following requirements:

   1. Neutrophil count ≥ 1 x 10^9/L, Hemoglobin ≥60g/L, platelets ≥ 50×109/L,
   2. Liver function: ALT ≤ 3 x ULN,AST≤3 x ULN, TBIL≤1.5 x ULN,
   3. Coagulation function: International standardized ratio (INR) ≤ 1.5x ULN, prothrombin time (PT) ≤1.5 x ULN,
   4. Cardiac function: good hemodynamic stability, left ventricular ejection fraction (LVEF) ≥55%.
4. Female subjects of childbearing potential and male subjects whose partner is a female of childbearing potential are required to use medically approved contraception or abstain from sex for at least 6 months during and at least 6 months after the end of the study treatment period; female subjects of childbearing potential have had a negative serum HCG test within 7 days prior to study enrollment and are not lactating;
5. Voluntarily participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

   Specific inclusion criteria:

   High-risk or relapsed/refractory primary membranous nephropathy
6. Primary membranous nephropathy diagnosed pathologically by renal biopsy;
7. Meets the clinical criteria for high-risk or recurrent/refractory membranous nephropathy, defined as:

   Subjects at risk who meet any of the following criteria: a) estimated glomerular filtration rate (eGFR, CKD-EPI equation) <60 mL/min/1.73m², and/or urine protein >8g/day persisting for more than 6 months;b) normal GFR, urinary protein >3.5 g/d, treated with ACEI/ARB for 6 months, urinary protein reduction <50%, and serum albumin <25 g/l or aPLA2R >50 RU/mL;

   Refractory membranous nephropathy subjects are defined as those who have shown poor response or resistance to previous immunosuppressive treatments (including corticosteroids and/or cytotoxic drugs, immunosuppressants and/or biologics), defined as persistent proteinuria ≥3.5g/day with a reduction of <50% compared to baseline;

   Recurrent membranous nephropathy is defined as a relapse (24-hour urinary protein ≥3.5 g) in subjects who have achieved complete or partial remission following treatment;
8. Subjects with relapsed/refractory MN and eGFR ≥ 45 mL/min/1.73 m2 during the screening period;
9. Primary IgA nephropathy pathologically confirmed by renal biopsy;
10. Subjects have medical records showing they have been on stable and maximally tolerated doses of either ACEI or ARB, as per local SOC and applicable guidelines, for at least 3 months preceding screening;
11. Subjects have been treated with hormones and/or cytotoxic drugs, immunosuppressants and/or biological agents (including but not limited to anti-CD20 monoclonal antibodies) for more than 6 months, and the 24-hour urine protein is ≥1.0 g; subjects with a rapidly progressive decline in kidney function (eGFR decreases by ≥50% within 3 months); or The subject relapsed after achieving complete remission/partial remission (CR/PR) following treatment (24-hour urine protein ≥1.0 g);
12. Estimated glomerular filtration rate (eGFR, CKD-EPI formula) ≥30 mL/min/1.73m2 at screening;
13. Meets the 2022 ACR/EULAR diagnostic criteria for ANCA-associated vasculitis, including microscopic polyangiitis, granulomatosis with polyangiitis, and eosinophilic granulomatosis with polyangiitis;
14. ANCA-related antibodies positive (MPO-ANCA or PR3-ANCA positive);
15. Kidney biopsy pathology is consistent with ANCA-associated vasculitis renal damage;
16. Birmingham Vasculitis Activity Score (BVAS) ≥15 points (total score 63 points), indicating active vasculitis;
17. At least two abnormalities related to the kidneys in the BVAS score;
18. Subjects meeting the definition of relapsed/refractory: standard treatment is ineffective or disease activity recurs after remission. Definition of conventional treatment: using glucocorticoids (more than 1mg/kg/day) and cyclophosphamide, along with any one of the following immunomodulatory drugs for ≥3 months: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biologics including rituximab, belimumab, and thalidomide;
19. Estimated glomerular filtration rate (eGFR, CKD-EPI formula) ≥30 mL/min/1.73m2 at screening

Exclusion Criteria:

Subjects who meet any of the following common exclusion criteria or disease-specific exclusion criteria will not be eligible for this study

Common exclusion Criteria:

1. Subjects known to have allergic reactions, hypersensitivity, intolerance, or contraindications to CD19/BCMA universal CAR-T or any drug components that may be used in the study (including fludarabine, cyclophosphamide, and tocilizumab), or who have previously experienced severe allergic reactions;
2. The subject has or is suspected of having uncontrolled or treatable fungal, bacterial, viral, or other infections;
3. Subjects with central nervous system disorders caused by autoimmune diseases or non-autoimmune diseases (including epilepsy, psychiatric disorders, organic brain syndrome, cerebrovascular accidents, encephalitis, central nervous system vasculitis);
4. Subjects with more serious heart conditions, such as angina, myocardial infarction, heart failure, and arrhythmias;
5. Subjects with congenital immunoglobulin deficiency;
6. The subject has other malignant tumours (excluding non-melanoma skin cancer and carcinoma in situ of the cervix, bladder cancer, and breast cancer with disease-free survival of over 5 years);
7. Subjects with end-stage renal failure;
8. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and have peripheral blood HBV DNA titres above the detection limit; subjects who are positive for hepatitis C virus (HCV) antibodies and peripheral blood HCV RNA; subjects who are positive for human immunodeficiency virus (HIV) antibodies; subjects who test positive for syphilis;
9. Subjects have mental illness and severe cognitive impairment;
10. Subjects who have participated in other clinical trials within 6 months prior to enrolment;
11. Female participants who are pregnant or planning to conceive;
12. Subjects with hypertension and diabetes uncontrolled by medication;
13. Researchers believe that there are other reasons why some subjects cannot be included in this study;

    Specific exclusion Criteria:

    Relapsed/Refractory Primary Membranous Nephropathy
14. Secondary membranous nephropathy (e.g., hepatitis B, systemic lupus erythematosus, drug-associated, malignancy-associated, etc.), or in combination with other renal diseases confirmed by renal biopsy;

    Relapsed/Refractory IgA Nephropathy
15. Exclude secondary IgA nephropathy, including but not limited to: anaphylactic purpura, ankylosing spondylitis, systemic lupus erythematosus, desiccation syndrome, viral hepatitis, cirrhosis of the liver, rheumatoid arthritis, and mixed connective tissue disease; or in combination with other renal diseases confirmed by renal biopsy;
16. Crescentic nephritis (pathologic diagnosis of >50% crescentic bodies), micrognathic nephropathy with IgA deposition, and other specific types of pathologic or clinical renal disease;

    Relapsed/refractory ANCA-associated vasculitis kidney damage
17. Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2;
18. If subjects have alveolar haemorrhage and requires invasive lung ventilation, the expected duration exceeds the screening time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | up to 52 weeks after infusion
  To characterize the safety of anti-CD19/BCMA U CAR T Cells (KN3601) for Relapsed/Refractory Immune Nephropathy
Incidence of Treatment Emergent Adverse Events (TEAEs) | up to 52 weeks after infusion
  To characterize the safety of anti-CD19/BCMA U CAR T Cells (KN3601) for Relapsed/Refractory Immune Nephropathy

SECONDARY OUTCOMES:
The overall response rate (ORR) | up to 52 weeks after infusion
  To characterize the efficacy of anti-CD19/BCMA U CAR T Cells for Relapsed/Refractory Immune Nephropathy
Disease control rate (DCR) | up to 52 weeks after infusion
  To characterize the efficacy of anti-CD19/BCMA U CAR T Cells for Relapsed/Refractory Immune Nephropathy
B cell depletion rate | up to 52 weeks after infusion
  To characterize the efficacy of anti-CD19/BCMA U CAR T Cells for Relapsed/Refractory Immune Nephropathy
B cell reconstitution | up to 52 weeks after infusion
  To characterize the efficacy of anti-CD19/BCMA U CAR T Cells for Relapsed/Refractory Immune Nephropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No